CLINICAL TRIAL: NCT01849991
Title: Safety and Effect of L. Reuteri on Biomarkers of Inflammation in Healthy Infants With Colic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, J. Marc Rhoads, Director, Pediatric Gastroentrologist, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-11-0203; HSC-MS-11-0203 (Other: University of Texas Health Science Center at Houston)
Record Dates: First submitted 2013-01-31; First posted 2013-05-09 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Gastrointestinal; Colic
Keywords: Crying; Fussiness; Gas; Hydrogen Breath; Fecal Calprotectin
MeSH Terms: conditions — Colic; Crying; Mucopolysaccharidosis IV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus reuteri (Active Comparator): The first arm of the cohort will include 30 patients on LR (5x10^8 cfu's orally once daily.)
  Interventions: Biological: Lactobacillus reuteri
- Sunflower Oil (Placebo Comparator): The second arm includes 15 subjects on placebo (sunflower oil.)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Lactobacillus reuteri — Lactobacillus reuteri oil drops are a natural product containing Lactobacillus reuteri (LR), which has traditionally been used for the establishment of a well-functioning gastrointestinal (GI) microbiota and prevention and treatment of mild diarrhea associated with GI-tract infections, travel or antibiotic treatment.
  The drug is a clear liquid when suspended in sunflower oil. The drug will be administered orally, 0.2cc once daily.
  Arms: Lactobacillus reuteri
Biological: Placebo — Placebo is sunflower oil (vehicle for LR). The placebo will be administered the same way as drug listed above.
  Arms: Sunflower Oil

SUMMARY:
This protocol is a study of the effects of Lactobacillus reuteri in 45 healthy infants with colic. The study is being conducted in order to prove treatment dose with probiotic (Lactobacillus reuteri) in a clinical setting is safe in healthy infants with colic.

DETAILED DESCRIPTION:
This study will evaluate the safety and tolerability of Lactobacillus reuteri in healthy infants with colic. Patients will be randomized to receive either L. reuteri at one dose orally for a total of 42 doses. The doses will be 5x108 (5 drops) during a satisfactory assessment of safety and tolerability. The time on study treatment is 6 months, and the target sample size is 45 healthy infants.

Secondly, the investigators aim to gather evidence supporting hypothesis of safety and tolerability of Lactobacillus reuteri by administering a physical examination and testing of complete blood count, liver tests, and serum electrolytes over a forty-two day period.

ELIGIBILITY:
Inclusion Criteria:

* Full-term babies with colic (21-90 days old, who cry/fuss > 3h daily x > 3d wk)
* baby must have more than 3h crying for enrollment

Exclusion Criteria:

* severe gastroesophageal reflux (throwing up or spitting up more than a teaspoon of milk > 8 times daily, projectile, bilious or bloody emesis)
* failure to thrive
* intrauterine growth retardation
* hematochezia (blood in the stools)
* diarrhea (watery stools that takes the shape of a container > 5x daily)
* fever (38.2 degrees)
* Premature infants (<37 wk gestation)

Ages: 3 Weeks to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2013-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
45 healthy infants with colic will receive LR (health-promoting bacteria) or placebo measuring any changes in their health status. | 92 days
  1. Physical Examination of infants will be performed to evaluate any adverse effects of LR.
  2. Electrolyte testing at baseline will evaluate for any inborn error of fluid and electrolyte balance and at end of treatment will evaluate for any adverse impact of LR in the subjects.

SECONDARY OUTCOMES:
Determine effect of L. reuteri in 45 infants with colic on gastrointestinal inflammation as assessed by fecal calprotectin. | 1, 42 & 92 days
  To examine for evidence of anti-inflammatory effects in the normal intestine, we will test fecal samples from all infants for calprotectin level.

OTHER OUTCOMES:
Measuring the change in crying times (Barr Diary) in 45 healthy infants with colic during the administration of L reuteri. | 92 days
  Clinical scoring of crying and fussing will be evaluated using the Barr diary which will show crying patterns.
Determine effects of L. reuteri in 45 healthy infants with colic measuring the immunologic responses with plasma cytokines and circulating regulatory T-cells. | 1& 42 days
  1. A panel of inflammatory biomarkers will be examined which includes Th1 cytokines (TNFα, IL-1β); a Th2 cytokine (IL-10), a cytokine which regulates maturation of Tregs (IL-2), a cytokine receptor (OPG), a marker of intestinal barrier function (TIMP-1) and a marker for autoimmunity (TWEAK). Biomarkers will be assessed by MSD human multiplex cytokine assays or R&D Human ELISA kit.
  2. We will determine if LR treatment affects the frequency of Tregs in PBMCs in normal babies with colic.
Determine effect of L. reuteri on gastrointestinal inflammation as assessed by fecal microbiota in 45 healthy infants with colic. | 1, 42 & 92 days
  A stool sample will be collected and analyzed to determine the effect on overall microbiota produced by the ingestion of LR.

CONTACTS AND LOCATIONS:
Overall Officials: J. Marc Rhoads, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Result] Fatheree NY, Liu Y, Taylor CM, Hoang TK, Cai C, Rahbar MH, Hessabi M, Ferris M, McMurtry V, Wong C, Vu T, Dancsak T, Wang T, Gleason W, Bandla V, Navarro F, Tran DQ, Rhoads JM. Lactobacillus reuteri for Infants with Colic: A Double-Blind, Placebo-Controlled, Randomized Clinical Trial. J Pediatr. 2017 Dec;191:170-178.e2. doi: 10.1016/j.jpeds.2017.07.036. Epub 2017 Sep 29. PMID 28969890
- [Derived] Rhoads JM, Collins J, Fatheree NY, Hashmi SS, Taylor CM, Luo M, Hoang TK, Gleason WA, Van Arsdall MR, Navarro F, Liu Y. Infant Colic Represents Gut Inflammation and Dysbiosis. J Pediatr. 2018 Dec;203:55-61.e3. doi: 10.1016/j.jpeds.2018.07.042. Epub 2018 Aug 31. PMID 30177353